CLINICAL TRIAL: NCT04491903
Title: REBOA for Out-of-hospital Cardiac Arrest
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn
Sponsor: neurescue (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SafeStudy2
Record Dates: First submitted 2020-07-22; First posted 2020-07-30 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REBOA (Experimental)
  Interventions: Procedure: REBOA

INTERVENTIONS:
Procedure: REBOA — Endovascular balloon occlusion of the aorta

SUMMARY:
Cardiac arrest is a major health problem that carries a high mortality rate. Substantial research and development have been put into changing the outcome of cardiac arrest and despite the advent of automated external defibrillators (AED), increase in bystander Cardiopulmonary resuscitation (CPR) and automated CPR devices (ACPR), the proportion of patient survival to hospital discharge has only minimally improved.

The objective is to investigate safety and performance of the Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) procedure as an adjunct to Advanced Life Support (ALS) for treatment of refractory cardiac arrest.

DETAILED DESCRIPTION:
The scope of the study is to collect data on patients with refractory out of hospital cardiac arrest (OHCA) for this feasibility study.

Data collected:

* from enrolment of the patient until hospital arrival
* every 24 hours
* at discharge or 7 days post enrollment
* at 30 days post enrollment

The investigation is initiated to investigate the safety and performance of the REBOA procedure for patients experiencing refractory OHCA.

ELIGIBILITY:
Inclusion Criteria:

* Witnessed cardiac arrest
* Bystander or professional CPR within 5 minutes
* Refractory cardiac arrest

Exclusion Criteria:

* End Tidal CO2 <1,3 kPa
* Traumatic cardiac arrest
* Women with known pregnancy
* Patients with known terminal disease
* Patients with known do-not-attempt-CPR order
* Patients with overdose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Central blood pressure | 1 hour

SECONDARY OUTCOMES:
Return of spontaneous circulation (ROSC) | 1 hour
Changes in cardiac rhythm following balloon inflation | 1 hour
During procedure - time from first needle stick to successful sheath insertion | 1 hour
During procedure - time from first needle stick to finalized balloon inflation | 1 hour
End-tidal CO2 (EtCO2) | 1 hour

IPD SHARING:
Plan to Share IPD: No
Individual request